CLINICAL TRIAL: NCT02020525
Title: The Impact of Lowering Transfusion Trigger on Patient Immune Response During Major Abdominal Surgery
Brief Title: Blood Transfusions and Immune Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Associate Professor in Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TRANSF-CYTOK
Record Dates: First submitted 2013-12-18; First posted 2013-12-25 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Infection After Transfusion; Transfusion-related Immunomodulation Reaction; Cytokine Storm; Surgery
MeSH Terms: conditions — Cytokine Release Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- restrictive transfusion strategy (Experimental): Patients allocated to the restrictive transfusion strategy were transfused only when their hemoglobin concentration decreased below 7.7 g d dL-1 and were then maintained at hemoglobin concentrations between 7.7 and 9.9 g d dL-1.
  Interventions: Procedure: restrictive transfusion strategy
- liberal transfusion strategy (Active Comparator): Patients assigned to the liberal strategy were transfused when their hemoglobin concentration fell below 9.9 g dL-1, aiming at maintaining hemoglobin at or above 10 g dL-1.
  Interventions: Procedure: liberal transfusion strategy

INTERVENTIONS:
Procedure: restrictive transfusion strategy — Patients allocated to the restrictive transfusion strategy were transfused only when their hemoglobin concentration decreased below 7.7 g d dL-1 and were then maintained at hemoglobin concentrations between 7.7 and 9.9 g d dL-1.
  Arms: restrictive transfusion strategy
Procedure: liberal transfusion strategy — Patients assigned to the liberal strategy were transfused when their hemoglobin concentration fell below 9.9 g dL-1, aiming at maintaining hemoglobin at or above 10 g dL-1.
  Arms: liberal transfusion strategy

SUMMARY:
* We have previously reported the results of the primary and secondary outcomes of a randomized study aiming to investigate the impact of a restrictive transfusion protocol on the magnitude of reduction in blood transfusion in a typically mixed general surgery population subjected to major abdominal surgery.
* The main finding of that study was a reduction in red blood cell usage with the implementation of a restrictive transfusion regimen. This was achieved without adversely affecting clinical outcome in the population studied.
* The aim of this secondary analysis performed on a subgroup of 20 patients from the original study was to determine whether there are any differences in the postoperative immunologic response, as expressed by the production of inflammatory mediators, between a restrictive approach to red cell transfusion and a more liberal strategy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, American Society of Anesthesiologists (ASA) distribution I-III, scheduled for elective upper major abdominal surgery

Exclusion Criteria:

* history of bleeding diathesis
* hereditary hemostatic defects such as hemophilias
* chronic anticoagulant administration
* refusal of transfusions for religious reasons
* ischemic heart disease (unstable angina or myocardial infarction within the last six months)
* preexisting infectious diseases
* preexisting autoimmune diseases
* use of corticosteroids or immunosuppressive drugs within the last six months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2004-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The number of units transfused per patient as well as the incidence of blood transfusions in each transfusion strategy group (restrictive versus liberal) | first five postoperative days

SECONDARY OUTCOMES:
time of initial mobilization postoperatively | first five postoperative days
time of first liquid food intake | first five postoperative days
time of first solid food intake | first five postoperative days
incidence of postoperative infectious complications | first five postoperative days

OTHER OUTCOMES:
Secondary post-hoc analysis performed on a subgroup of 20 patients from the original study in order to determine whether there are any differences in the postoperative immunologic response between the two transfusion allocation groups | preoperatively, six, 24 and 72 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DEAA, Principal Investigator — Aretaieion University Hospital
Locations (1):
- Aretaieion University Hospital, Athens, Greece

REFERENCES:
- [Background] Baigrie RJ, Lamont PM, Kwiatkowski D, Dallman MJ, Morris PJ. Systemic cytokine response after major surgery. Br J Surg. 1992 Aug;79(8):757-60. doi: 10.1002/bjs.1800790813. PMID 1393463
- [Background] Koch CG, Li L, Sessler DI, Figueroa P, Hoeltge GA, Mihaljevic T, Blackstone EH. Duration of red-cell storage and complications after cardiac surgery. N Engl J Med. 2008 Mar 20;358(12):1229-39. doi: 10.1056/NEJMoa070403. PMID 18354101
- [Background] Vamvakas EC, Blajchman MA. Deleterious clinical effects of transfusion-associated immunomodulation: fact or fiction? Blood. 2001 Mar 1;97(5):1180-95. doi: 10.1182/blood.v97.5.1180. No abstract available. PMID 11222359
- [Background] Leal Noval SR, Jara Lopez I. Do multiple blood transfusions predispose for a higher rate of non-blood-related infection complications? Clin Microbiol Infect. 2002 Jul;8(7):383-7. doi: 10.1046/j.1469-0691.2002.00465.x. PMID 12199847
- [Background] Hebert PC, Wells G, Blajchman MA, Marshall J, Martin C, Pagliarello G, Tweeddale M, Schweitzer I, Yetisir E. A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. N Engl J Med. 1999 Feb 11;340(6):409-17. doi: 10.1056/NEJM199902113400601. PMID 9971864
- [Background] Sherry RM, Cue JI, Goddard JK, Parramore JB, DiPiro JT. Interleukin-10 is associated with the development of sepsis in trauma patients. J Trauma. 1996 Apr;40(4):613-6; discussion 616-7. doi: 10.1097/00005373-199604000-00016. PMID 8614042
- [Background] Bilgin YM, Brand A. Transfusion-related immunomodulation: a second hit in an inflammatory cascade? Vox Sang. 2008 Nov;95(4):261-71. doi: 10.1111/j.1423-0410.2008.01100.x. PMID 19138255
- [Result] Theodoraki K, Markatou M, Rizos D, Fassoulaki A. The impact of two different transfusion strategies on patient immune response during major abdominal surgery: a preliminary report. J Immunol Res. 2014;2014:945829. doi: 10.1155/2014/945829. Epub 2014 Apr 3. PMID 24804272